CLINICAL TRIAL: NCT03846427
Title: A Phase 2, Open-label Study of Zanubrutinib (BGB-3111) in Patients With Relapsed or Refractory Marginal Zone Lymphoma
Brief Title: Study of Zanubrutinib (BGB-3111) in Participants With Marginal Zone Lymphoma
Acronym: MAGNOLIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-214; 2018-001284-24 (EudraCT Number); CTR20180823 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2018-10-11; First posted 2019-02-19 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Marginal Zone Lymphoma; MZL
Keywords: BGB-3111; Zanubrutinib
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Zanubrutinib 160 mg (two 80-mg capsules) orally twice daily with or without food until progressive disease, intolerable toxicity, or withdrawal of consent
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib at a dose of 160 mg orally twice a day (BID)
  Other Names: BGB-3111; Brukinsa

SUMMARY:
This is a single arm study to evaluate the efficacy, safety and tolerability of zanubrutinib (BGB-3111) in participants with relapsed/refractory marginal zone lymphoma (R/R MZL).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18 years or older
2. Histologically confirmed diagnosis of MZL including splenic, nodal, and extranodal subtypes
3. Previously received one or more lines of therapy including at least one CD20-directed regimen (either as monotherapy or as chemoimmunotherapy) with documented failure to achieve at least partial response or documented progressive disease (PD) after, the most recent systemic treatment
4. Current need for systemic therapy for MZL
5. Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI)
6. Eastern Cooperative Oncology Group (ECOG) of 0-2
7. Life expectancy ≥ 6 months
8. Adequate bone marrow function
9. Adequate organ function
10. Male and female participants must use highly effective methods of contraception

Key Exclusion Criteria:

1. Known transformation to aggressive lymphoma, eg, large cell lymphoma
2. Clinically significant cardiovascular disease
3. Prior malignancy within the past 2 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer
4. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
5. History of stroke or intracranial hemorrhage
6. Severe or debilitating pulmonary disease
7. Active fungal, bacterial and/or viral infection requiring systemic therapy
8. Known central nervous system involvement by lymphoma
9. Known infection with HIV, or serologic status reflecting active viral hepatitis B (HBV) or viral hepatitis C (HCV) infection
10. Major surgery within 4 weeks of the first dose of study drug
11. Prior treatment with a Bruton's tyrosine kinase (BTK) inhibitor
12. Pregnant or lactating women
13. Requires ongoing treatment with a strong Cytochrome P4503A (CYP3A) inhibitor or inducer
14. Concurrent participation in another therapeutic clinical trial

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (31):
- United States (2):
  - Clinical Research Alliance, Inc, Westbury, New York
  - The Charlotte Mecklenburg Hospital Authority, Charlotte, North Carolina
- Australia (8):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - The Saint George Hospital Kogarah, Kogarah, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Bedford PK, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- University Hospital Vinohrady Hematology Department, Prague, Czechia
- France (4):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Hopital de La Conception Aphm, Marseille
  - Hopital Saint Louis, Paris
  - Chu Hopital Lyon Sud, PierreBenite
- Italy (5):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Universita Degli Studi Di Modena Azienda Ospedaliere Policlinco, Modena
  - Azienda Ospedaliera S Maria Di Terni, Terni
  - Ao Citta Della Salute E Della Scienza Di Torino Presidio O, Torino
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Takapuna
- Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi, South Korea
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie Hospital, Greater Manchester
  - University College Hospital, London
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Stephen Opat, Robert Marcus, MA, FRCP, FRCPath, Craig A. Portell, MD, William Reed, MD, Chris Tankersley, Jane Huang, MD, Judith Trotman, MBChB, FRACP, FRCPA. Phase 2 Study of Zanubrutinib (BGB-3111) in Patients with Relapsed/Refractory Marginal Zone Lymphoma. Blood. 2019; 134(1):5256. https://doi.org/10.1182/blood-2019-122629
- [Background] Stephen Opat, et al. Efficacy and Safety of Zanubrutinib in Patients with Relapsed/Refractory Marginal Zone Lymphoma: Initial Results of the MAGNOLIA (BGB-3111-214) Trial. Presented at the 62nd American Society of Hematology (ASH) Annual Meeting, December 5-8, 2020. Abstract 339.
- [Background] Opat S, Tedeschi A, Linton K, McKay P, Hu B, Chan H, Jin J, Sobieraj-Teague M, Zinzani PL, Coleman M, Thieblemont C, Browett P, Ke X, Sun M, Marcus R, Portell CA, Ardeshna K, Bijou F, Walker P, Hawkes EA, Mapp S, Ho SJ, Talaulikar D, Zhou KS, Co M, Li X, Zhou W, Cappellini M, Tankersley C, Huang J, Trotman J. The MAGNOLIA Trial: Zanubrutinib, a Next-Generation Bruton Tyrosine Kinase Inhibitor, Demonstrates Safety and Efficacy in Relapsed/Refractory Marginal Zone Lymphoma. Clin Cancer Res. 2021 Dec 1;27(23):6323-6332. doi: 10.1158/1078-0432.CCR-21-1704. Epub 2021 Sep 15. PMID 34526366
- [Background] Opat S, Tedeschi A, Hu B, et al: Long-term efficacy and safety of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma. 2022 ASH Annual Meeting and Exposition. Abstract 234. Presented December 10, 2022.
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Opat S, Tedeschi A, Hu B, Linton KM, McKay P, Leitch S, Coleman M, Zinzani PL, Jin J, Sun M, Sobieraj-Teague M, Browett P, Ke X, Thieblemont C, Ardeshna K, Bijou F, Walker P, Hawkes EA, Ho SJ, Zhou K, Liang Z, Xu J, Tankersley C, Delarue R, Co M, Trotman J. Safety and efficacy of zanubrutinib in relapsed/refractory marginal zone lymphoma: final analysis of the MAGNOLIA study. Blood Adv. 2023 Nov 28;7(22):6801-6811. doi: 10.1182/bloodadvances.2023010668. PMID 37682792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 31 study centers in 9 countries.
Pre-assignment Details: The study was composed of an initial screening phase (up to 35 days), a single-arm treatment phase, and a follow-up phase. A total of 38 participants rolled over to BGB-3111-LTE1 (NCT04170283) after study completion.
Period: Overall Study
Arm/Group | Zanubrutinib
Started | 68
Completed | 51
Not Completed | 17
Not completed — Death | 13
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.9 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13
  White | 40
  Multiple | 2
  Other | 1
  Unknown | 1
  Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Independent Review Committee (IRC) Assessment
Description: ORR is defined as the percentage of participants with complete or partial response as the best overall response, as determined by an IRC using the Lugano Classification
Time Frame: Up to approximately 3 years and 2.5 months
Population: Efficacy analysis set consisted of all participants with a confirmed diagnosis of MZL who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 68.2 [55.56 to 79.11]
Statistical Analysis 1: Comparison: Zanubrutinib; Test type: Superiority — P value was based on the exact binomial test against the null hypothesis of ORR = 30% with alternative of ORR > 30%; p < 0.0001, Binomial exact method

2. Secondary Outcome: ORR by Investigator Assessment
Description: ORR is defined as the percentage of participants with complete or partial response as the best overall response, as determined by the investigator using the Lugano Classification.
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 75.8 [63.64 to 85.46]

3. Secondary Outcome: ORR by IRC Assessment Using Positron Emission Tomography-Computed Tomography (PET-CT)
Description: ORR is defined as the percentage of participants with complete and partial response as the best overall response, as determined by an IRC using PET-CT assessment data for participants with fluorodeoxyglucose (FDG)-avid disease
Time Frame: Up to approximately 3 years and 2.5 months
Population: Efficacy analysis set consisted of evaluable participants with FDG-avid disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 59
Percentage of participants | 69.5 [56.13 to 80.81]

4. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the investigator using Lugano Classification
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Months | NA [16.5 to NA] — Not estimable due to insufficient number of participants with events

5. Secondary Outcome: PFS Event-Free Rate by Investigator Assessment
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the investigator using Lugano Classification. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for PFS at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 57.9 [44.83 to 68.86]

6. Secondary Outcome: PFS by IRC Assessment
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by an IRC using Lugano Classification
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Months | NA [27.6 to NA] — Not estimable due to insufficient number of participants with events

7. Secondary Outcome: PFS Event-Free Rate by IRC Assessment
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the IRC using Lugano Classification. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for PFS at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 70.9 [57.20 to 80.95]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first study drug administration to the date of death due to any cause
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Months | NA [NA to NA] — Not estimable due to insufficient number of participants with events

9. Secondary Outcome: OS Event-Free Rate
Description: OS is defined as the time from first study drug administration to the date of death due to any cause. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for OS at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 85.9 [74.7 to 92.4]

10. Secondary Outcome: Duration of Response (DOR) by Investigator Assessment
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the investigator using Lugano Classification.
Time Frame: Up to approximately 3 years and 2.5 months
Population: Efficacy analysis set consisted of all participants with a confirmed diagnosis of MZL who received at least 1 dose of study drug; DOR was summarized for responders only, defined as participants with a best overall response of partial response or above.
Measure: Median (Full Range); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 50
Months | NA [22.1 to NA] — Not estimable due to insufficient number of participants with events

11. Secondary Outcome: DOR Event-Free Rate by Investigator Assessment
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the investigator using Lugano Classification. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for progression or death at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 50
Percentage of participants | 60.8 [44.8 to 73.6]

12. Secondary Outcome: DOR by IRC Assessment
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the IRC using Lugano Classification.
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 10
Measure: Median (Full Range); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 45
Months | NA [25.0 to NA] — Not estimable due to insufficient number of participants with events

13. Secondary Outcome: DOR Event-Free Rate by IRC Assessment
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the IRC using Lugano Classification. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for progression or death at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 45
Percentage of participants | 72.9 [54.4 to 84.9]

14. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from study treatment start to the date of discontinuation of study drug due to any reason.
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Months | 27.8 [14.7 to NA] — Not estimable due to insufficient number of participants with events and high censoring rate for time-to-event variable

15. Secondary Outcome: TTF Event-Free Rate
Description: TTF is defined as the time from study treatment start to the date of discontinuation of study drug due to any reason. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for TTF at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 53.0 [40.4 to 64.2]

16. Secondary Outcome: Time to Next Line of Therapy
Description: Time to next line of therapy is defined as the time from study treatment start to the start of the first subsequent therapy for MZL
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Months | NA [NA to NA] — Not estimable due to insufficient number of participants with events

17. Secondary Outcome: Time to Next Line of Therapy Event-Free Rate
Description: Time to next line of therapy is defined as the time from study treatment start to the start of the first subsequent therapy for MZL. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for time to next line of therapy at 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: Up to 3 years and 2.5 months after first participant enrolled; Month 24 reported
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Percentage of participants | 74.5 [61.7 to 83.6]

18. Secondary Outcome: Time to Response (TTR) by Investigator Assessment
Description: TTR is defined as the time from study treatment start to date of the earliest qualifying response (partial response or better) as assessed by the investigator using Lugano Classification
Time Frame: Up to approximately 3 years and 2.5 months
Population: Efficacy analysis set consisted of all participants with a confirmed diagnosis of MZL who received at least 1 dose of study drug; TTR was summarized for responders only, defined as participants with a best overall response of partial response or above.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 50
Months | 2.79 [1.7 to 16.6]

19. Secondary Outcome: TTR by IRC Assessment
Description: TTR is defined as the time from study treatment start to date of the earliest qualifying response (partial response or better), as assessed by the IRC using Lugano Classification.
Time Frame: Up to approximately 3 years and 2.5 months
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 45
Months | 2.79 [1.7 to 11.1]

20. Secondary Outcome: Change From Baseline in EuroQol 5-dimension 5-level (EQ-5D-5L) Visual Analogue Score (VAS)
Description: Mean change from baseline in EQ-5D-5L VAS. The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' Positive change from baseline indicates improved health.
Time Frame: Baseline to Cycle 30 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Score on a scale
  Cycle 3: number analyzed (Participants) | 57
  Cycle 3 | 1.0 (18.18)
  Cycle 6: number analyzed (Participants) | 50
  Cycle 6 | 2.2 (15.78)
  Cycle 9: number analyzed (Participants) | 47
  Cycle 9 | 0.2 (16.28)
  Cycle 12: number analyzed (Participants) | 42
  Cycle 12 | 2.8 (16.15)
  Cycle 18: number analyzed (Participants) | 33
  Cycle 18 | 5.6 (17.68)
  Cycle 24: number analyzed (Participants) | 35
  Cycle 24 | 5.8 (15.24)
  Cycle 30: number analyzed (Participants) | 28
  Cycle 30 | 1.6 (18.15)

21. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status
Description: Mean change from baseline in EORTC QLQ-C30 Global Health Status/Quality of Life score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of cancer patients and includes global health status and quality of life questions related to their overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Answers are converted to a score of 0 to 100, with a positive score from baseline indicating improved health.
Time Frame: Baseline to Cycle 30 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 66
Score on a scale
  Cycle 3: number analyzed (Participants) | 58
  Cycle 3 | 7.471 (19.5396)
  Cycle 6: number analyzed (Participants) | 49
  Cycle 6 | 7.823 (15.8121)
  Cycle 9: number analyzed (Participants) | 48
  Cycle 9 | 5.382 (20.0833)
  Cycle 12: number analyzed (Participants) | 42
  Cycle 12 | 7.143 (17.3216)
  Cycle 18: number analyzed (Participants) | 32
  Cycle 18 | 10.677 (18.4811)
  Cycle 24: number analyzed (Participants) | 35
  Cycle 24 | 9.286 (19.2561)
  Cycle 30: number analyzed (Participants) | 28
  Cycle 30 | 6.250 (20.4910)

22. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory tests, physical exams, and vital signs
Time Frame: From first dose to 30 days after last dose of study drug (Up to approximately 3 years and 2.5 months)
Population: Safety analysis set is all participants who were enrolled and received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 68
Participants
  At least one TEAE | 68
  At least one SAE | 30

23. Secondary Outcome: Area Under the Curve From Time 0 to 6 Hours (AUC0-6)
Time Frame: Predose (within 30 min prior to dose) and 0.5, 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 (28 days per cycle)
Population: Pharmacokinetic analysis set included all participants who had at least 1 postdose zanubrutinib plasma concentration
Measure: Mean (Standard Deviation); unit: Hour*ng/mL
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 9
Hour*ng/mL | 868.0 (304.3)

24. Secondary Outcome: Apparent Oral Clearance (CL/F) of Zanubrutinib
Time Frame: Predose (within 30 min prior to dose) and 0.5, 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 (28 days per cycle)
Population: Pharmacokinetic analysis set included all participants who had at least 1 postdose zanubrutinib plasma concentration
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 8
Liters/hour | 215.3 (114.8)

25. Secondary Outcome: Maximum Observed Concentration (Cmax)
Time Frame: Predose (within 30 min prior to dose) and 0.5, 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 (28 days per cycle)
Population: Pharmacokinetic analysis set included all participants who had at least 1 postdose zanubrutinib plasma concentration
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 11
nanograms/milliliter | 315.5 (120.2)

26. Secondary Outcome: Elimination Half Life (t1/2)
Time Frame: Predose (within 30 min prior to dose) and 0.5, 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 (28 days per cycle)
Population: Pharmacokinetic analysis set included all participants who had at least 1 postdose zanubrutinib plasma concentration
Measure: Median (Full Range); unit: Hours
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 9
Hours | 1.2 [0.8 to 2.7]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose of study drug (Up to approximately 3 years and 2.5 months)
Description: Defined as an adverse event that had an onset date or worsening in severity from baseline on or after the date of first dose of study drug up to 30 days after study drug discontinuation or initiation of new anticancer therapy, whichever occurred first.
Arm/Group | Zanubrutinib
All-Cause Mortality (participants affected / at risk) | 13/68
Serious Adverse Events (participants affected / at risk) | 30/68
Other Adverse Events (participants affected / at risk) | 61/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=68)
Anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Pyrexia (General disorders) | 3
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Septic encephalopathy (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar infarction (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=68)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 6
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 8
COVID-19 (Infections and infestations) | 6
Oral herpes (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 16
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 4
Weight decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03846427/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03846427/SAP_001.pdf